CLINICAL TRIAL: NCT04650555
Title: A Phase 1 Dose Escalation Trial Evaluating the Safety and Pharmacokinetic Profile of BIO 300 Oral Powder in Healthy Volunteers
Brief Title: BIO 300 Oral Powder Safety and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanetics Corporation (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); Joint Warfighter Medical Research Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CL0106-01
Record Dates: First submitted 2020-11-19; First posted 2020-12-02 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Acute Radiation Syndrome
MeSH Terms: conditions — Acute Radiation Syndrome | interventions — Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single Ascending Dose Cohort 1 (Experimental): 500 mg BIO 300 Oral Powder administered as a single dose
  Interventions: Drug: BIO 300 Oral Powder
- Single Ascending Dose Cohort 2 (Experimental): 1000 mg BIO 300 Oral Powder, if dose escalation criteria met, administered as a single dose
  Interventions: Drug: BIO 300 Oral Powder
- Single Ascending Dose Cohort 3 (Experimental): 2000 mg BIO 300 Oral Powder, if dose escalation criteria met, administered as a single dose
  Interventions: Drug: BIO 300 Oral Powder
- Single Ascending Dose Cohort 4 (Experimental): Single dose to be determined based on the safety and pharmacokinetic profiles in cohorts 1-3
  Interventions: Drug: BIO 300 Oral Powder
- Multiple Single Dose Cohort 5 (Experimental): Highest dose or maximum tolerated dose from the Single Ascending Dose study administered as a single dose given daily for 6 consecutive days
  Interventions: Drug: BIO 300 Oral Powder

INTERVENTIONS:
Drug: BIO 300 Oral Powder — Amorphous solid dispersion of genistein milled into a powder
  Other Names: BIO 300; Genistein

SUMMARY:
Open-label, single ascending dose and multiple single dose study in healthy volunteers to evaluate the safety and pharmacokinetics of BIO 300 Oral Powder (BIO 300). The single ascending dose study consists of 4 ascending dose cohorts and the multiple single dose study consists of a single dose given daily for 6 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult non-smokers, 18-64 years old.
2. BMI 18-32 kg/m^2.
3. No ingestion of prescription or over-the-counter medications (including dietary and herbal supplements) for 7 days prior to first dose of study drug and no planned use during study participation. Acetaminophen of up to 3 g/day and ibuprofen up to 1 g/day will be allowed at discretion of the Investigator.
4. At the discretion of the Investigator, blood routine, liver and kidney functions are within the controllable range.

   1. Adequate hepatic function as evidenced by ALT, AST or LDH < 1.25X ULN and bilirubin < 1.5X ULN for the reference lab.
   2. Adequate renal function as evidenced by a serum creatinine ≤ 1.5 X ULN for the reference laboratory OR a calculated creatinine clearance of ≥ 60 mL/min by the Cockcroft-Gault Equation.
   3. Adequate hematopoietic function as evidenced by white blood cells ≥ 3x10^9 / L and platelets ≥ 100x10^9 / L.
5. Female subjects of childbearing potential must have a negative pregnancy test within 72 hours of the start of treatment.
6. Subjects must agree to abstain from heterosexual intercourse or use a reliable method of contraception for 7 days after their last dose. Subjects using hormonal contraception are required to utilize condom/spermicide + additional barrier method for 7 days after their last dose.
7. Ability to read and provide written informed consent.
8. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, dietary restrictions, and other study procedures.
9. No clinically significant abnormalities identified by medical history, physical examination, vital signs, ECG, and clinical laboratory tests in the opinion of the Investigator.

Exclusion Criteria:

1. Any prior use of the study test article.
2. Any clinically significant weight loss any time in prior 4 weeks at discretion of Investigator based on medical history interview.
3. Subjects with any of the following are not eligible;

   1. Previous history of QTc prolongation resulting from "known-risk" medications (www.Crediblemeds.org) that required discontinuation of that medication;
   2. Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age;
   3. Presence of left bundle branch block (LBBB);
   4. QTc with Fridericia's correction (QTcF) that is unmeasurable, or ≥ 480 msec on screening ECG. The average QTcF from the screening ECG (completed in triplicate) must be < 480 msec in order for the subject to be eligible for the study.
4. Subjects must not have had a clinically significant cardiac event such as myocardial infarction (within 6 months prior to the first dose of the study treatment); uncontrolled/symptomatic congestive heart failure (New York Heart Association (NYHA) classification of heart disease, Class III or IV, see Appendix 3) within 6 months before entry; or the presence of any other uncontrolled cardiovascular conditions [unstable hypertension at discretion of Investigator or arrhythmia, unstable angina pectoris, or severe valvular heart disease, etc.] that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
5. Subjects with a history of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE Grade 3) or asymptomatic sustained ventricular tachycardia are not eligible. Subjects with atrial fibrillation with well-controlled ventricular rate are eligible at the discretion of the Investigator.
6. Psychiatric conditions, social situations or substance abuse that precludes the ability of the subject to cooperate with the requirements of the trial and protocol therapy at Investigator discretion.
7. Inability to refrain from alcohol consumption for 48 hours prior to day 1 and for the duration of the study. Illicit drugs, including THC, must be avoided from screen through the duration of the study.
8. Grade 2 or higher peripheral neuropathy.
9. Positive results for Hep B surface antigen, Hep C antibody, or HIV 1/2 antibody at screening visit.
10. Clinically significant immunodeficiency disorder in the opinion of the Investigator.
11. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
12. Women who are breastfeeding are not eligible for this study.
13. Subjects that are vegan, vegetarian or consume a soy-rich diet.
14. Any history of systemic infection requiring hospitalization, systemic antibiotics, or as judged clinically significant by the investigator in the 3 months prior to day 1.
15. Any condition possibly affecting drug absorption (e.g., prior bariatric surgery, gastrectomy, intestinal resection). Participants who have undergone appendectomy or cholecystectomy are allowed so long as the surgery occurred more than 6 months prior to day 1.
16. Treatment with another investigational drug within 30 days or 5 half-lives (whichever is longer) proceeding Day 1.
17. Positive drug screen or alcohol test at screen and day 1 predose.
18. Blood donation of approximately 1 pint (500 ml) or more within 60 days of day 1; plasma donations within 14 days of day 1. Subjects must agree not to donate blood or plasma for the duration of the study and for 30 days following end of study procedures.
19. Inability to swallow powdered medication followed with water.
20. History of sensitivity to heparin or heparin-induced thrombocytopenia.
21. Considered by the Investigator to be unsuitable to participate in the study for any other reason.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Kaytor, Ph.D., Principal Investigator — Humanetics Corporation
Locations (1):
- Nucleus Network, Ltd (Formally Prism Research, LLC), Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Serebrenik AA, Verduyn CW, Kaytor MD. Safety, Pharmacokinetics, and Biomarkers of an Amorphous Solid Dispersion of Genistein, a Radioprotectant, in Healthy Volunteers. Clin Pharmacol Drug Dev. 2023 Feb;12(2):190-201. doi: 10.1002/cpdd.1188. Epub 2022 Oct 27. PMID 36301689

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Ascending Dose Cohort 1 | Single Ascending Dose Cohort 2 | Single Ascending Dose Cohort 3 | Single Ascending Dose Cohort 4 | Multiple Single Dose Cohort 5
Started | 6 | 6 | 6 | 6 | 10
Completed | 6 | 6 | 5 | 6 | 8
Not Completed | 0 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Ascending Dose Cohort 1 | Single Ascending Dose Cohort 2 | Single Ascending Dose Cohort 3 | Single Ascending Dose Cohort 4 | Multiple Single Dose Cohort 5 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 10 | 34
Age, Continuous [Median (Full Range); unit: years] | 55 [27 to 59] | 37 [28 to 58] | 40 [22 to 62] | 48 [19 to 63] | 46 [22 to 65] | 45 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 3 | 5 | 18
  Male | 2 | 3 | 3 | 3 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 6 | 6 | 10 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 2
  White | 5 | 6 | 5 | 5 | 8 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 10 | 34

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Related to BIO 300 Oral Powder
Description: Evaluate the safety of single and multiple dose BIO 300 Oral Powder administration
Time Frame: Day 1 up to 1 week for Single Ascending Dose and Day 1 up to 2 weeks for Multiple Single Dose
Population: No adverse events were reported for the Single Ascending Dose Cohort 1
Measure: Number; unit: Number of Adverse Events
Units Other Than Participants: Number of Adverse Events
Arm/Group | Single Ascending Dose Cohort 1 | Single Ascending Dose Cohort 2 | Single Ascending Dose Cohort 3 | Single Ascending Dose Cohort 4 | Multiple Single Dose Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 10
Number analyzed (Number of Adverse Events) | 0 | 5 | 4 | 6 | 26
Number of Adverse Events
  Dose Limiting Toxicities |  | 0 | 0 | 0 | 0
  Unlikely Treatment-Related Adverse Events |  | 1 | 0 | 0 | 2
  Possibly Treatment-Related Adverse Events |  | 0 | 0 | 3 | 7
  Probably Treatment-Related Adverse Events |  | 4 | 4 | 0 | 15
  Definitely Treatment-Related Adverse Events |  | 0 | 0 | 2 | 1
  Unrelated Adverse Event |  | 0 | 0 | 1 | 1

2. Primary Outcome: Change in ECG QTc Interval
Description: Measurement of the average QTc interval with Fridericia's correction (completed in triplicate at each timepoint)
Time Frame: Day 1 up to 1 week after the last dose for Single Ascending Dose and Multiple Single Dose Cohorts
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Single Ascending Dose Cohort 1 | Single Ascending Dose Cohort 2 | Single Ascending Dose Cohort 3 | Single Ascending Dose Cohort 4 | Multiple Single Dose Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 10
milliseconds
  Screening | 407 (9.3) | 402 (19.3) | 416 (21.8) | 415 (18.7) | 413 (13.3)
  4 Hours Post First Dose | 412 (9.6) | 407 (16.5) | 419 (27.8) | 420 (16.3) | 417 (7.4)
  24 Hours Post First Dose | 407 (11.3) | 400 (11.2) | 402 (26.7) | 404 (41.7) | 413 (9.9)
  1 Week Post Last Dose | 408 (12.4) | 401 (18.3) | 416 (36.3) | 414 (12.6) | 415 (9.0)

3. Primary Outcome: Change in Clinical Laboratory Values
Description: Monitoring of blood serum levels of albumin and total protein (all reported as g/dL)
Time Frame: Day 3 and 7 for Single Ascending Dose and Day 3, 6 and 13 for Multiple Single Dose
Population: Participants in the single ascending dose study were assessed on days 3 and 7 and participants in the multiple dose study were assessed on days 3, 6 and 13
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Single Ascending Dose Cohort 1 | Single Ascending Dose Cohort 2 | Single Ascending Dose Cohort 3 | Single Ascending Dose Cohort 4 | Multiple Single Dose Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
g/dL
  Albumin Day 3 | 4.483 (0.204) | 4.433 (0.393) | 4.333 (0.367) | 4.550 (0.187) | 4.225 (0.349)
  Albumin Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Albumin Day 6 |  |  |  |  | 4.475 (0.249)
  Albumin Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Albumin Day 7 | 4.233 (0.216) | 4.283 (0.279) | 4.440 (0.241) | 4.517 (0.117) |
  Albumin Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Albumin Day 13 |  |  |  |  | 4.475 (0.306)
  Total Protein Day 3 | 6.667 (0.344) | 6.833 (0.638) | 6.500 (0.369) | 6.650 (0.547) | 6.363 (0.444)
  Total Protein Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Total Protein Day 6 |  |  |  |  | 6.788 (0.348)
  Total Protein Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Total Protein Day 7 | 6.417 (0.331) | 6.850 (0.619) | 6.520 (0.438) | 6.717 (0.454) |
  Total Protein Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Total Protein Day 13 |  |  |  |  | 6.550 (0.518)

4. Primary Outcome: Change in Clinical Laboratory Values
Description: Monitoring of blood serum levels of bicarbonate, chloride, potassium, and sodium (all reported as mEq/L)
Time Frame: Day 3 and 7 for Single Ascending Dose and Day 3, 6 and 13 for Multiple Single Dose
Population: Analyzed on Day 3 and 7 for Single Ascending Dose and Day 3, 6 and 13 for Multiple Single Dose
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Single Ascending Dose Cohort 1 | Single Ascending Dose Cohort 2 | Single Ascending Dose Cohort 3 | Single Ascending Dose Cohort 4 | Multiple Single Dose Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
mEq/L
  Bicarbonate Day 3 | 26.833 (1.722) | 26.167 (0.753) | 27.167 (2.401) | 27.500 (1.049) | 23.875 (2.850)
  Bicarbonate Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Bicarbonate Day 6 |  |  |  |  | 23.750 (1.165)
  Bicarbonate Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Bicarbonate Day 7 | 26.500 (1.871) | 27.500 (1.761) | 29.000 (0.707) | 28.667 (1.751) |
  Bicarbonate Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Bicarbonate Day 13 |  |  |  |  | 23.125 (1.246)
  Chloride Day 3 | 104.5 (2.429) | 104.0 (1.549) | 104.7 (0.816) | 103.5 (0.837) | 105.5 (1.927)
  Chloride Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Chloride Day 6 |  |  |  |  | 103.8 (2.252)
  Chloride Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Chloride Day 7 | 104.3 (1.366) | 104.5 (1.761) | 104.2 (1.095) | 104.8 (2.317) |
  Chloride Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Chloride Day 13 |  |  |  |  | 105.1 (0.835)
  Potassium Day 3 | 4.417 (0.271) | 4.500 (0.141) | 4.617 (0.306) | 4.400 (0.303) | 4.288 (0.318)
  Potassium Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Potassium Day 6 |  |  |  |  | 4.413 (0.336)
  Potassium Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Potassium Day 7 | 4.217 (0.279) | 4.483 (0.306) | 4.580 (0.460) | 4.233 (0.151) |
  Potassium Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Potassium Day 13 |  |  |  |  | 4.288 (0.155)
  Sodium Day 3 | 140.7 (1.966) | 139.5 (1.225) | 140.7 (0.816) | 140.2 (1.835) | 140.0 (1.414)
  Sodium Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Sodium Day 6 |  |  |  |  | 139.5 (1.414)
  Sodium Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Sodium Day 7 | 140.0 (1.265) | 139.2 (1.472) | 139.2 (1.304) | 142.3 (2.066) |
  Sodium Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Sodium Day 13 |  |  |  |  | 140.1 (1.727)

5. Primary Outcome: Change in Clinical Laboratory Values
Description: Monitoring of blood serum levels of bilirubin (total and direct), BUN, calcium, cholesterol (total), creatinine, HDL, glucose, magnesium, phosphorous, triglycerides, and uric acid (all reported as mg/dL)
Time Frame: Day 3 and 7 for Single Ascending Dose and Day 3, 6 and 13 for Multiple Single Dose
Population: Analyzed Day 3 and 7 for Single Ascending Dose and Day 3, 6 and 13 for Multiple Single Dose
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Single Ascending Dose Cohort 1 | Single Ascending Dose Cohort 2 | Single Ascending Dose Cohort 3 | Single Ascending Dose Cohort 4 | Multiple Single Dose Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
mg/dL
  Total Bilirubin Day 3 | 0.467 (0.308) | 0.417 (0.117) | 0.333 (0.137) | 0.650 (0.501) | 0.613 (0.394)
  Total Bilirubin Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Total Bilirubin Day 6 |  |  |  |  | 0.500 (0.185)
  Total Bilirubin Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Total Bilirubin Day 7 | 0.483 (0.331) | 0.583 (0.417) | 0.340 (0.167) | 0.400 (0.141) |
  Total Bilirubin Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Total Bilirubin Day 13 |  |  |  |  | 0.563 (0.307)
  Direct Bilirubin Day 3 | 0.200 (0) | 0.200 (0) | 0.200 (0) | 0.200 (0) | 0.200 (0)
  Direct Bilirubin Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Direct Bilirubin Day 6 |  |  |  |  | 0.200 (0)
  Direct Bilirubin Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Direct Bilirubin Day 7 | 0.200 (0) | 0.200 (0) | 0.200 (0) | 0.200 (0) |
  Direct Bilirubin Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Direct Bilirubin Day 13 |  |  |  |  | 0.200 (0)
  BUN Day 3 | 18.00 (3.46) | 13.33 (2.94) | 14.83 (4.62) | 13.50 (4.51) | 11.88 (3.09)
  BUN Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  BUN Day 6 |  |  |  |  | 12.00 (2.83)
  BUN Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  BUN Day 7 | 16.67 (4.23) | 14.50 (2.88) | 14.20 (5.85) | 13.83 (4.26) |
  BUN Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  BUN Day 13 |  |  |  |  | 11.63 (3.82)
  Calcium Day 3 | 9.73 (0.37) | 9.38 (0.32) | 9.27 (0.23) | 9.72 (0.33) | 9.25 (0.34)
  Calcium Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Calcium Day 6 |  |  |  |  | 9.60 (0.19)
  Calcium Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Calcium Day 7 | 9.47 (0.14) | 9.37 (0.26) | 9.18 (0.37) | 9.50 (0.32) |
  Calcium Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Calcium Day 13 |  |  |  |  | 9.36 (0.30)
  Cholesterol Day 3 | 200 (43) | 181 (23) | 158 (19) | 210 (44) | 178 (23)
  Cholesterol Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Cholesterol Day 6 |  |  |  |  | 193 (22)
  Cholesterol Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Cholesterol Day 7 | 195 (34) | 180 (33) | 173 (32) | 213 (49) |
  Cholesterol Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Cholesterol Day 13 |  |  |  |  | 177 (26)
  Creatinine Day 3 | 0.905 (0.182) | 0.943 (0.154) | 0.883 (0.180) | 0.900 (0.127) | 0.944 (0.116)
  Creatinine Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Creatinine Day 6 |  |  |  |  | 1.030 (0.099)
  Creatinine Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Creatinine Day 7 | 0.873 (0.147) | 1.028 (0.150) | 0.954 (0.212) | 0.980 (0.131) |
  Creatinine Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Creatinine Day 13 |  |  |  |  | 1.043 (0.094)
  HDL Day 3 | 52 (11) | 55 (15) | 52 (10) | 69 (21) | 49 (14)
  HDL Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  HDL Day 6 |  |  |  |  | 55 (15)
  HDL Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  HDL Day 7 | 52 (9) | 54 (16) | 56 (9) | 71 (23) |
  HDL Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  HDL Day 13 |  |  |  |  | 52 (17)
  Glucose Day 3 | 95.2 (8.0) | 89.7 (7.3) | 90.7 (6.5) | 90.2 (8.8) | 96.3 (5.8)
  Glucose Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Glucose Day 6 |  |  |  |  | 93.6 (5.2)
  Glucose Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Glucose Day 7 | 101.5 (10.0) | 92.3 (2.7) | 97.0 (12.1) | 105.8 (40.8) |
  Glucose Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Glucose Day 13 |  |  |  |  | 93.4 (4.7)
  Magnesium Day 3 | 2.10 (0.11) | 2.05 (0.14) | 2.07 (0.12) | 1.90 (0.17) | 1.98 (0.10)
  Magnesium Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Magnesium Day 6 |  |  |  |  | 2.05 (0.17)
  Magnesium Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Magnesium Day 7 | 2.02 (0.12) | 2.12 (0.10) | 2.06 (0.11) | 1.98 (0.12) |
  Magnesium Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Magnesium Day 13 |  |  |  |  | 2.06 (0.09)
  Phosphorous Day 3 | 3.58 (0.37) | 3.62 (0.45) | 3.75 (0.41) | 3.52 (0.34) | 3.14 (0.36)
  Phosphorous Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Phosphorous Day 6 |  |  |  |  | 3.49 (0.34)
  Phosphorous Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Phosphorous Day 7 | 3.62 (0.53) | 3.68 (0.42) | 3.70 (0.49) | 3.68 (0.62) |
  Phosphorous Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Phosphorous Day 13 |  |  |  |  | 0.39 (0.54)
  Triglycerides Day 3 | 80.2 (43.3) | 104.2 (91.0) | 80.5 (37.5) | 85.5 (30.6) | 101.9 (38.8)
  Triglycerides Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Triglycerides Day 6 |  |  |  |  | 98.6 (23.3)
  Triglycerides Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Triglycerides Day 7 | 71.3 (22.1) | 117.3 (107.0) | 79.2 (44.5) | 80.5 (39.7) |
  Triglycerides Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Triglycerides Day 13 |  |  |  |  | 89.8 (20.6)
  Uric Acid Day 3 | 5.25 (1.08) | 4.62 (1.26) | 4.48 (1.16) | 5.07 (1.38) | 5.20 (1.50)
  Uric Acid Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Uric Acid Day 6 |  |  |  |  | 5.21 (1.55)
  Uric Acid Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Uric Acid Day 7 | 5.13 (1.09) | 5.30 (1.89) | 4.10 (0.73) | 5.08 (1.24) |
  Uric Acid Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Uric Acid Day 13 |  |  |  |  | 5.20 (1.60)

6. Primary Outcome: Change in Clinical Laboratory Values
Description: Monitoring of blood serum levels of alkaline phosphatase, ALT, amylase, AST, LDH, and lipase (all reported as IU/L)
Time Frame: Day 3 and 7 for Single Ascending Dose and Day 3, 6 and 13 for Multiple Single Dose
Population: Analyzed day 3 and 7 for Single Ascending Dose and Day 3, 6 and 13 for Multiple Single Dose
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Single Ascending Dose Cohort 1 | Single Ascending Dose Cohort 2 | Single Ascending Dose Cohort 3 | Single Ascending Dose Cohort 4 | Multiple Single Dose Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
IU/L
  ALP Day 3 | 74.2 (18.1) | 66.7 (13.9) | 64.2 (18.8) | 62.8 (21.4) | 59.5 (15.5)
  ALP Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  ALP Day 6 |  |  |  |  | 60.3 (16.2)
  ALP Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  ALP Day 7 | 69.5 (14.7) | 69.0 (17.3) | 68.0 (21.1) | 52.5 (29.7) |
  ALP Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  ALP Day 13 |  |  |  |  | 59.4 (18.6)
  ALT Day 3 | 18.2 (5.7) | 21.2 (18.6) | 15.2 (3.2) | 16.2 (9.5) | 17.6 (5.5)
  ALT Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  ALT Day 6 |  |  |  |  | 18.4 (4.1)
  ALT Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  ALT Day 7 | 16.7 (3.9) | 27.8 (24.1) | 17.8 (6.3) | 16.7 (10.7) |
  ALT Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  ALT Day 13 |  |  |  |  | 18.1 (5.1)
  Amylase Day 3 | 26.5 (8.0) | 32.2 (13.7) | 21.8 (8.7) | 26.8 (8.0) | 28.0 (7.9)
  Amylase Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Amylase Day 6 |  |  |  |  | 32.8 (10.1)
  Amylase Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Amylase Day 7 | 25.8 (7.3) | 30.3 (13.4) | 22.6 (10.1) | 26.8 (10.5) |
  Amylase Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Amylase Day 13 |  |  |  |  | 29.8 (8.8)
  AST Day 3 | 19.0 (3.6) | 19.7 (6.0) | 21.2 (6.4) | 21.8 (6.1) | 17.8 (3.7)
  AST Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  AST Day 6 |  |  |  |  | 19.6 (4.3)
  AST Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  AST Day 7 | 19.2 (3.7) | 26.3 (11.9) | 23.6 (10.9) | 22.2 (6.1) |
  AST Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  AST Day 13 |  |  |  |  | 18.1 (5.1)
  LDH Day 3 | 170 (20) | 147 (14) | 152 (31) | 171 (48) | 158 (15)
  LDH Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  LDH Day 6 |  |  |  |  | 166 (19)
  LDH Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  LDH Day 7 | 171 (22) | 157 (27) | 161 (17) | 179 (39) |
  LDH Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  LDH Day 13 |  |  |  |  | 173 (21)
  Lipase Day 3 | 26.2 (4.9) | 42.8 (31.9) | 23.8 (10.7) | 33.3 (10.6) | 28.6 (8.4)
  Lipase Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Lipase Day 6 |  |  |  |  | 35.5 (13.6)
  Lipase Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6 | 0
  Lipase Day 7 | 26.8 (3.9) | 35.8 (10.5) | 26.6 (13.6) | 32.0 (13.3) |
  Lipase Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8
  Lipase Day 13 |  |  |  |  | 31.4 (9.3)

7. Primary Outcome: Area Under Curve of Genistein-Aglycone in Serum
Description: Area under the curve of BIO 300 Oral Powder as assessed by analyzing serum concentrations of genistein-aglycone (free genistein) at multiple timepoints
Time Frame: Day 1 for the Single Ascending Dose and Day 6 for the Multiple Single Dose, prior to 1st dose then 0.5, 1, 2, 4, 6, 8, 12, 24, and 48 hours post dose and Day 1 Multiple Single Dose prior to dosing then 0.5, 1, 2, and 4 hours post dose
Population: Area under the curve from 0 to 48 hours (AUC 0-48)
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Arm/Group | Single Ascending Dose Cohort 1 | Single Ascending Dose Cohort 2 | Single Ascending Dose Cohort 3 | Single Ascending Dose Cohort 4 | Multiple Single Dose Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
ng/mL*hr | 902.9 (605.1) | 1530.9 (518.2) | 1730.8 (361.6) | 5836.0 (3280.8) | 2957.3 (1222.4)

8. Secondary Outcome: Number of Differentially Expressed Genes From Whole Blood Samples
Description: The number of significantly differentially expressed genes detected in whole blood samples at various timepoints after BIO 300 Oral Powder dosing. Significant differential gene expression was defined as genes that have a mean absolute log2 fold change >2 with an adjusted p-value of <0.05 relative to baseline expression levels.
Time Frame: Day 1 for the Single Ascending Dose prior to dosing then 1, 2, 4, and 24 hours post dose and Day 1 Multiple Single Dose prior to dosing then 1, 2, and 4 hours post dose and and Day 6 prior to dosing then 4, 8, 12 and 24 hours post dose
Population: All participants had samples collected for RNA sequencing. Overall number of participants analyzed indicates the number of participants from each cohort that had samples analyzed by RNA sequencing.
Measure: Number; unit: Differentially expressed genes
Arm/Group | Single Ascending Dose Cohort 1 | Single Ascending Dose Cohort 2 | Single Ascending Dose Cohort 3 | Single Ascending Dose Cohort 4 | Multiple Single Dose Cohort 5
Number analyzed (Participants) | 4 | 0 | 4 | 4 | 7
Differentially expressed genes
  Day 1, 1 hr post-dose | 0 |  | 0 | 0 | 0
  Day 1, 2 hr post-dose | 0 |  | 0 | 0 | 0
  Day 1, 4 hr post-dose | 0 |  | 1 | 0 | 0
  Day 1, 24 hr post-dose | 0 |  | 0 | 0 | 0
  Day 6, 4 hr post-dose | 0 |  | 0 | 0 | 0
  Day 6, 8 hr post-dose | 0 |  | 0 | 0 | 6
  Day 6, 12 hr post-dose | 0 |  | 0 | 0 | 7
  Day 6, 24 hr post-dose | 0 |  | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening to 1 week after the last dose of BIO 300 Oral Powder (up to 5 weeks)
Arm/Group | Single Ascending Dose Cohort 1 | Single Ascending Dose Cohort 2 | Single Ascending Dose Cohort 3 | Single Ascending Dose Cohort 4 | Multiple Single Dose Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 0/6 | 4/6 | 2/6 | 5/6 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Ascending Dose Cohort 1 (N=6) | Single Ascending Dose Cohort 2 (N=6) | Single Ascending Dose Cohort 3 (N=6) | Single Ascending Dose Cohort 4 (N=6) | Multiple Single Dose Cohort 5 (N=10)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (6)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Lipase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 4 (4)
Lightheaded (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perioral Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT04650555/Prot_SAP_000.pdf